CLINICAL TRIAL: NCT06963164
Title: Feasibility of a Remotely-Delivered, Technology-Enabled, Joint Protection Program
Brief Title: Testing of a New Joint Protection Program
Acronym: "Helping Hand"
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: The Arthritis Society, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15417
Record Dates: First submitted 2025-03-27; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-03

CONDITIONS: Hand Osteoarthritis
Keywords: hand osteoarthritis; randomize controlled trial; feasibility; pilot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Joint Protection Program (Experimental): The content will be organised into 6 modules (4 asynchronous, 2 live modules). Each module will focus on specific principles or activities.
  The first two modules will present general information on Hand Osteoarthritis and Joint Protection Principles, and the third module will be activity-based and will go through different tasks including Activities of Daily Living, Occupational Activities, Household Chores, Hobbies, and Various Functional Everyday Activities. The fourth module will be pre-recorded, and it will include a patient partner talking about their experiences living with hand osteoarthritis.
  The two live modules will happen bi-weekly interchangeably. The first module will be a community of practice, where people will get together and exchange information on tools, strategies, and resources for hand osteoarthritis. The second module will include open Q&A sessions, where patients will get the chance to talk to a clinician and ask questions about managing hand osteoarthritis.
  Interventions: Other: Helping Hand - Joint Protection Program
- Waitlist (No Intervention): The participants in this group will continue to receive Standard Care and they will be offered access to the program after the end of the 12 weeks.

INTERVENTIONS:
Other: Helping Hand - Joint Protection Program — Joint protection refers to a set of techniques and strategies that help reduce stress on the joints, manage pain, and prevent further joint damage. These techniques are particularly important for people with hand arthritis, as the small joints in the hands are often affected, leading to pain, stiffness, and difficulty performing daily tasks. Key principles of joint protection include:
  1. Using larger, stronger joints whenever possible (e.g., using the forearm instead of the fingers to push open a door).
  2. Reducing strain by spreading the load across multiple joints (e.g., carrying items with two hands instead of one).
  3. Avoid tight gripping or pinching motions that can overstrain the joints.
  4. Incorporating assistive devices to reduce effort during tasks (e.g., jar openers or ergonomic tools).
  5. Pacing and prioritizing activities to avoid overuse of the joints and allow for adequate rest
  Arms: Joint Protection Program

SUMMARY:
The goal of this study is to to examine the feasibility of a full-scale trial on Helping Hand, a new Joint Protection Program for Hand Osteoarthritis and to examine the acceptability of the new Joint Protection Program.

This study will not assess the effectiveness of the program, as it is not designed or powered to do so. Instead, the information gathered will be used to refine the trial design and ensure the future full-scale trial that will assess the effectiveness of the program is robust and successful. The acceptability of the new Joint Protection Program will be assessed through a survey that will be administered to the intervention group at the end of the trial, which will be based on a standardized acceptability framework

Participants will:

Gain access to an online Joint Protection Program or continue to receive usual care for 12 weeks Visit the clinic or complete online assessments once every 4 weeks Keep a diary of their symptoms and the number of times they used other interventions to manage their symptoms (i.e. painkillers)

DETAILED DESCRIPTION:
The goal of this study is to to examine the feasibility of a definite trial on Helping Hand, a new Joint Protection Program for Hand Osteoarthritis and to examine the acceptability of the new Joint Protection Program.

Joint protection refers to a set of techniques and strategies that help reduce stress on the joints, manage pain, and prevent further joint damage. These techniques are particularly important for people with hand arthritis, as the small joints in the hands are often affected, leading to pain, stiffness, and difficulty performing daily tasks. Key principles of joint protection include:

1. Using larger, stronger joints whenever possible (e.g., using the forearm instead of the fingers to push open a door).
2. Reducing strain by spreading the load across multiple joints (e.g., carrying items with two hands instead of one).
3. Avoid tight gripping or pinching motions that can overstrain the joints.
4. Incorporating assistive devices to reduce effort during tasks (e.g., jar openers or ergonomic tools).
5. Pacing and prioritizing activities to avoid overuse of the joints and allow for adequate rest.

By adopting these strategies, people with hand arthritis can minimize discomfort and preserve their ability to perform daily activities. This research is important because hand arthritis can make everyday tasks-like opening jars, getting dressed, or gardening-painful and difficult. Current resources for managing arthritis often lack a focus on practical, evidence-based strategies tailored to the needs of people with hand arthritis.

This feasibility study will test the practicality of running a future full-scale randomized controlled trial and the acceptability of the intervention. The feasibility testing includes evaluating key trial processes such as recruitment rates (how many people agree to participate), randomization (how well participants are assigned to groups), attrition rates (how many people stay in the study until the end), adherence (whether participants follow the program as intended), and clinical outcome completion rates (how many participants complete the required assessments). The acceptability of the intervention will be assessed through a survey that will be administered to the intervention group at the end of the trial, which will be based on a standardized acceptability framework. Importantly, this study will not assess the effectiveness of the program, as it is not designed or powered to do so. Instead, the information gathered will be used to refine the trial design and ensure the future full-scale trial is robust and successful.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of hand osteoarthritis Pain symptoms for at least 3 months Ability to use a smartphone, tablet, or computer Ability to communicate in English

Exclusion Criteria:

Presence of neurological disorders, dementia, or other cognitive conditions that could interfere with trial procedures Scheduled hand surgery within the next 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rates | 4, 8, and 12-weeks after randomization
  Pre-defined cut-off scores will be used. Based on the cut-off scores each outcome will be categorised in one of three categories: "proceed"; "proceed with modifications"; and "do not proceed". Recruitment rates will be classified as proceed if they achieve or surpass the predefined threshold set at 8-10 participants on average per month.
Adherence | 4, 8, and 12-weeks after randomization
  Uptake/participation will be tracked electronically by recording when participants log onto the website and monitoring whether participants show up in the live sessions. Adherence will also be measured by having the participants track the weekly modifications they performed through a self-reported diary. Pre-defined cut-off scores will be used. Based on the cut-off scores each outcome will be categorised in one of three categories: "proceed"; "proceed with modifications"; and "do not proceed". Adherence to the intervention protocol will be categorized as "proceed" if it achieves a minimum adherence rate of 85%.
Clinical outcome measure completion | baseline, 4, 8, and 12-weeks after randomization
  Pre-defined cut-off scores will be used. Based on the cut-off scores each outcome will be categorised in one of three categories: "proceed"; "proceed with modifications"; and "do not proceed". Outcome completeness will be considered "proceed" when data collection for at least 90% of the intended outcomes is achieved.
Attrition Rates | 4, 8, and 12-weeks after randomization
  Pre-defined cut-off scores will be used. Based on the cut-off scores each outcome will be categorised in one of three categories: "proceed"; "proceed with modifications"; and "do not proceed". Attrition rates will be classified as "proceed" if they remain below the predefined threshold, typically set at 20% or lower

CONTACTS AND LOCATIONS:
Locations (1):
- Roth | McFarlane Hand and Upper Limb Centre (HULC), London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No